CLINICAL TRIAL: NCT07036757
Title: PROJECT EATT: Enjoying Affordable and Tasty Food Together
Brief Title: Enjoying Affordable and Tasty Food Together
Acronym: PROJECT EATT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: BJ's Wholesale Club (Unknown)
Responsible Party: Principal Investigator, Sabrina Noel, Associate Professor, University of Massachusetts, Lowell
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#24
Record Dates: First submitted 2025-05-07; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Food Insecurity; Dietary Quality; Quality of Life; Cooking Self-efficacy; Perceived Stress; Anxiety; Depressive Symptomatology; Anthropometrics: Height and Weight; Glucose Variability; Blood Pressure
Keywords: Nutrition Education; Cardiometabolic outcomes; Meal Kits; Stress and Mental Health; Quality of Life
MeSH Terms: conditions — Anxiety Disorders; Body Weight; Psychological Well-Being | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal Kit and Nutrition Education arm (Experimental): Receives the meal kit intervention and nutrition education education materials.
  Interventions: Other: Meal Kit and Nutrition Education
- Usual care (No Intervention): Receives standard of care, which will include printed materials from the Dietary Guidelines for Americans on eating a healthy diet and complementary recipes.

INTERVENTIONS:
Other: Meal Kit and Nutrition Education — Meal kits contain ingredients for 3 meals designed for 4 servings, along with nutrition education materials, recipes, and information on how to store and prepare the meals. Weekly educational content focused on healthy eating, food security, and meal planning will be provided, either via print materials or through an online platform (e.g., email or app-based resources).
  Arms: Meal Kit and Nutrition Education arm

SUMMARY:
The goal of this pilot study is to examine the feasibility of a novel meal kit and nutrition education intervention among adults aged 40 years and older, who are lower income, and to evaluate the preliminary impact of the meal kit and nutrition education intervention on food insecurity, dietary quality, mental health, quality of life and cardiovascular risk factors compared with general nutrition education materials in this population.

The main questions are:

What is the acceptability and satisfaction with the meal kits and nutrition education intervention?

What are the participation rates in the nutrition education program and the evaluation of the intervention?

What is the impact of the intervention on food insecurity, dietary quality and cooking and food preparation self-efficacy compared with general nutrition education materials?

What is the impact of the intervention of psychosocial health, quality of life and cardiometabolic outcomes compared with general nutrition education materials?

DETAILED DESCRIPTION:
Food insecurity is a major risk factor for chronic health conditions through mechanisms such as poorer dietary quality and higher intake of processed foods due to high cost of healthier foods, poorer psychosocial health from increased stress and depression due to the worry of not having enough food, tradeoffs in spending and priorities to purchase food, and increased immune system activation and inflammation. Individuals who have lower income reported barriers to healthy eating beyond just access to healthy foods, including lack of time to prepare meals, insufficient nutrition knowledge, and limited cooking skills. Programs that reduce burden related to shopping, planning, and cooking time, and that do not solely provide food, may be more successful in reducing food insecurity and increasing dietary quality long term. Pre-made meals (ready to eat), tailored for specific diseases, have been shown to be beneficial for people living with health outcomes like diabetes. While pre-made meals designed for specific diseases can improve health outcomes,19-21 they do not address nutrition knowledge and cooking efficacy, which are important for developing long term behavior change. Meal kits are a growing area of food retail because they reduce challenges with meal planning and grocery shopping, but the majority of studies that have examined meal kits in relation to outcomes do not include nutrition education, particularly focused on cultural relevance.

The proposed pilot study is a randomized trial to evaluate the feasibility and whether a meal kit and nutrition education program leads to greater improvements in food insecurity, dietary quality, cooking and food preparation self-efficacy, psychosocial outcomes, quality of life, and cardiometabolic outcomes (glucose variability, blood pressure and anthropometric measures) compared with printed nutrition education materials and complementary recipes.

After successful screening and consent, 120 participants will be randomly assigned to either:

Group 1 (Intervention group, n=60): Receives the meal kit intervention and nutrition education weekly for 12 weeks. The meal kits, which include all ingredients needed to make a meal and step-by-step instructions for making the meal, will be delivered to participants homes. Participants will received meal kits to make 3 meals per week containing up to 4-5 servings for families.

Group 2 (Control group, n=60): Receives standard of care, which will include printed materials on eating a healthy diet and complementary recipes weekly.

Assessments will occur at baseline and 12-week follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years and older.
* Household income at or less than the 200% the federal poverty level (household size 1: $30,120, household size 2: $40,880, household size 3: $51,640, household size 4: $62,400, and household size 5: $73,160)
* Willing to provide informed consent and complete the study requirements, including attending study visits and completing questionnaires.
* Access to a refrigerator or other means to safely store perishable food, as the meal kits require refrigeration.
* BMI > 30 kg/m2 and self-report having at least one of the following: elevated blood pressure or hypertension, elevated glucose, prediabetes or diabetes.
* Reside in the Greater Lowell area or surrounding regions to ensure feasibility of meal kit delivery and data collection.

Exclusion Criteria:

* Less than 40 years old
* Does not have BMI >30 kg/m2, elevated blood pressure or hypertension, or elevated glucose, prediabetes or diabetes
* Not able to provide consent (adults lacking capacity)
* Follow a medically restricted diet or have allergies to wheat, soy, or dairy
* Plans to move from the Greater Lowell area within the next 12 months
* Live outside the Greater Lowell area because this will impact meal kit delivery
* Individuals without a working refrigerator in your household
* Have a serious medical condition requiring a doctor's care including cancer, chronic kidney disease and/or celiac disease
* Currently part of a study on diabetes, cardiovascular disease, nutrition or weight-loss
* Currently taking any weight loss medication like Ozempic, or medication for diabetes, dyslipidemia or hypertension
* Currently using a continuous glucose monitor

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-28 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Food insecurity | At enrollment and at 12 weeks
  The U.S. Department of Agriculture (USDA) 10-item food security screener will be used. This tool asks participants about their food security within the last 12 months. Scores range from 0 to 10, which a score of 0 indicating high food security, 1-2 indicating marginal food security, 3-5 indicating low food security, and 6-10 indicating very low food security.
Dietary Quality | At enrollment and at 12 weeks
  Dietary data will be collected by three 24-hr dietary recalls, using multi-pass interview software. At each time point, one 24-hour recall will be conducted during the interview, and two by phone within the following week (including a weekend day). A trained interviewer will use the Nutrition Data System for Research software (NDSR version 2019; Nutrition Coordinating Center, University of Minnesota).
Perceived Stress | At enrollment and at 12 weeks
  Perceived Stress Scale: The 14- item Perceived Stress Scale (PSS) gauges the respondent's perception of stress over the last month. The PSS measures the extent to which respondents perceive their lives over the past month as unpredictable and uncontrollable. Total scores ranges from 0-56, with higher scores indicating greater perceived stress.
Anxiety | At enrollment and at 12 weeks
  The State Trait Anxiety Scale assesses anxiety in participants using a 10-item questionnaire. Total scores range from 10 to 40, with greater scores indicating greater anxiety symptoms.
Depressive Symptomatology | At enrollment and at 12 weeks
  The Center for Epidemiological Studies Depression Scale (CES-D) will be used to assess depressive symptomatology. The scale consists of 20 items which ask about mood during the past week. Total scores range from 0 to 60, with higher scores indicating more severe depressive symptomatology.
Health-related Quality of Life | At enrollment and at 12 weeks
  Health-related QOL will be assessed using the validated U.S. Centers for Disease Control and Prevention (CDC) Health-Related Quality of Life (HRQOL) scale. This instrument includes the standard 4-item set of Healthy Days core questions. Scores range from 0 to 30 days with higher scores indicating more frequent poor physical and mental health.
Blood Pressure | At enrollment and at 12 weeks
  Systolic and diastolic blood pressure will be measured using an electronic sphygmomanometer (DinamapTM Model 8260, Critikon, Tampa, FL), in duplicate, after a short rest period.
Body Mass Index | At enrollment and at 12 weeks
  Height and weight will be measured in duplicate following standard techniques and integrated into one reported measures of body mass index. Weight will be measured with a clinical scale (Toledo Weight Plate, Model I5S, Bay State and Systems Inc. Burlington, MA), and height with a portable stadiometer. Body mass index (BMI, kg/m2) will be calculated as weight in kilograms divided by height in meters squared.
Glucose variability | At enrollment and at 12 weeks
  Interstitial glucose will be measured every 15 minutes using Dexcom G6 PRO continuous glucose monitors. Monitors will be fitted by trained research study staff on the upper, non-dominant arm with adhesive tape during the baseline visit and work for 7 days. The monitor will be removed by trained staff.
Waist circumference | At enrollment and 12 weeks.
  Waist circumference will be measured in duplicate using a flexible tape measure following standard procedures. An average of the two values will be used.

IPD SHARING:
Plan to Share IPD: No